CLINICAL TRIAL: NCT02978261
Title: A Phase I, Open-label, Dose Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics (PK) of PLB1001 in Patients With PTPRZ1-MET Fusion Gene Positive Recurrent High-grade Gliomas
Brief Title: Study of a c-Met Inhibitor PLB1001 in Patients With PTPRZ1-MET Fusion Gene Positive Recurrent High-grade Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Pearl Biotechnology Limited Liability Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMO-PLB1001-I-GBM-01
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2018-08

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PLB1001 (Experimental): There are 4 dose cohorts, including 50mg BID,100mg BID, 200mg BID and 300mg BID in the dose escalation stage and PLB1001 will be administered orally to patients twice daily for each dose cohort.
  Interventions: Drug: PLB1001

INTERVENTIONS:
Drug: PLB1001 — PLB1001 is a capsule in the form of 25 mg and 100mg, twice daily.
  Other Names: Bozitinib

SUMMARY:
This phase I, open-label, dose-escalation study was conducted to determine the maximum tolerated dose (MTD), recommended phase II dose (RP2D), dose-limiting toxicities (DLTs), pharmacokinetics (PK) profile, and preliminary antitumor activity of single and multiple doses of PLB1001 in Patients with PTPRZ1-MET fusion gene positive recurrent high-grade Gliomas.

DETAILED DESCRIPTION:
This is a Phase I, open-label study of PLB1001 administered orally to patients with PTPRZ1-MET fusion gene positive recurrent high-grade Gliomas. The aim of dose-escalation study is to estimate the MTD and to identify the dose-limiting toxicity(DLT) and the recommended phase II dose (RP2D) for PLB1001 single agent as well as to determine the PK/PD profile. Aprox. 20 patients will be enrolled in this study.

PLB1001 is a potent selective c-Met inhibitor. PLB1001 acts on cancer by blocking abnormal cMET-mediated signaling (including PTPRZ1-MET fusion gene), leading to profound tumor growth inhibition in xenografts of PTPRZ1-MET fusion gene positive glioblastoma tumor.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age≥18 years
* Histologically or cytologically confirmed recurrent high-grade glioma after concurrent or adjuvant chemoradiotherapy
* Prior treatment with temozolomide
* Must have evidence of PTPRZ1-MET fusion gene positivity from the results of molecular pre-screening evaluations
* At least one measurable lesion as per RANO
* No evidence of recent haemorrhage on baseline MRI of the brain
* Stable or decreasing dose of corticosteroids within 5 days prior to the first dose
* Major surgery within 4 weeks prior to first dose of PLB1001
* Previous anti-cancer and investigational agents within 4 weeks before first dose of PLB1001. If previous treatment is a monoclonal antibody, then the treatment must be discontinued at least 6 weeks before first dose of PLB1001
* Pregnant or nursing women
* Involved in other clinical trials <30 days prior to first dose
* Prior therapy with gamma knife or other focal high-dose radiotherapy is allowed, but the patient must have subsequent histologic documentation of recurrence, unless the recurrence is a new lesion outside the irradiated field
* Karnofsky performance status ≥ 50%

Exclusion Criteria:

* Previous or current treatment with a c-Met inhibitor or HGF-targeting therapy
* The subject is unable to undergo MRI scan (e.g. has pacemaker)
* Clinically significant, uncontrolled heart diseases： Unstable angina; History of documented congestive heart failure (New York Heart Association functional classification> II); Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 145 mm Hg and/or Diastolic Blood Pressure (DBP) ≥85 mm Hg; Arrhythmias.
* Active peptic ulcer disease or gastritis
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 1, except for alopecia
* Major surgery within 4 weeks prior to first dose of PLB1001
* Previous anti-cancer and investigational agents within 4 weeks before first dose of PLB1001. If previous treatment is a monoclonal antibody, then the treatment must be discontinued at least 6 weeks before first dose of PLB1001
* Pregnant or nursing women
* Involved in other clinical trials <30 days prior to first dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with dose-limiting toxicities | 2 years
  The primary endpoint is evaluation of safety and tolerability during all the study of therapy following the initiation of single and multiple doses of PLB1001. The safety and tolerability variables to be evaluated in this study are adverse events, vital signs, and electrocardiograms (ECGs), Incidence and nature of DLTs (Dose-Limiting Toxicities), to determine the MTD (Maximum Tolerated Dose).

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of PLB1001 and its metabolite | Day 1-3 Single Dose and Day 1-28 Steady State
  In the study of single-dose, full Pharmacokinetics(PK) profiles of PLB1001 will be obtained following administration of a single oral dose of PLB1001 on Day 1 to Day 2. At multiple-dose, Pharmacokinetics(PK) sampling will include a pre-dose and at the 0.5, 1, 2, 4, 6, 8, 10, 12, 14 and 16 hour time points on days 1and 15 of dosing in the first 28-Day cycle of therapy, and pre-dose on days 2, 16 and 17 of the first 28-Day cycle of therapy
Maximum plasma concentration observed (Cmax) of PLB1001 and its metabolite | Day 1-3 Single Dose and Day 1-28 Steady State
  In the study of single-dose, full Pharmacokinetics(PK) profiles of PLB1001 will be obtained following administration of a single oral dose of PLB1001 on Day 1 to Day 2. At multiple-dose, Pharmacokinetics(PK) sampling will include a pre-dose and at the 0.5, 1, 2, 4, 6, 8, 10, 12, 14 and 16 hour time points on days 1and 15 of dosing in the first 28-Day cycle of therapy, and pre-dose on days 2, 16 and 17 of the first 28-Day cycle of therapy
Time to Cmax (Tmax) of PLB1001 and its metabolite | Day 1-3 Single Dose and Day 1-28 Steady State
  In the study of single-dose, full Pharmacokinetics(PK) profiles of PLB1001 will be obtained following administration of a single oral dose of PLB1001 on Day 1 to Day 2. At multiple-dose, Pharmacokinetics(PK) sampling will include a pre-dose and at the 0.5, 1, 2, 4, 6, 8, 10, 12, 14 and 16 hour time points on days 1and 15 of dosing in the first 28-Day cycle of therapy, and pre-dose on days 2, 16 and 17 of the first 28-Day cycle of therapy
Preliminary antitumor activity of PLB1001 | 2 years
  Preliminary antitumor activity of PLB1001 assessed using RANO

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Li, MD, Principal Investigator — Beijing Shijitan Hospital, CMU
Locations (1):
- Beijing Shijitan Hospital,CMU, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hu H, Mu Q, Bao Z, Chen Y, Liu Y, Chen J, Wang K, Wang Z, Nam Y, Jiang B, Sa JK, Cho HJ, Her NG, Zhang C, Zhao Z, Zhang Y, Zeng F, Wu F, Kang X, Liu Y, Qian Z, Wang Z, Huang R, Wang Q, Zhang W, Qiu X, Li W, Nam DH, Fan X, Wang J, Jiang T. Mutational Landscape of Secondary Glioblastoma Guides MET-Targeted Trial in Brain Tumor. Cell. 2018 Nov 29;175(6):1665-1678.e18. doi: 10.1016/j.cell.2018.09.038. Epub 2018 Oct 18. PMID 30343896